CLINICAL TRIAL: NCT03733899
Title: An Investigation of the Impact of Localized Topical Anesthesia of the Ocular Surface on End-of-day Contact Lens Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6292
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Results first posted 2020-02-06 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Upper lid margin/Lower lid margin/Cornea (Experimental): Subjects that are at least 18 years of age wearing their habitual lenses will be randomized into one of six unique sequences of an ocular surface region. For each region within a sequence, the two treatments will be randomly assigned to the left and right eye (anesthesia left eye/placebo right eye OR placebo left eye/anesthesia left eye).
  Interventions: Diagnostic Test: Local Anesthesia; Diagnostic Test: Placebo
- Lower lid margin/Cornea/ Upper lid margin (Experimental): Subjects that are at least 18 years of age wearing their habitual lenses will be randomized into one of six unique sequences. For each region within a sequence, the two treatments will be randomly assigned to the left and right eye (anesthesia left eye/placebo right eye OR placebo left eye/anesthesia left eye).
  Interventions: Diagnostic Test: Local Anesthesia; Diagnostic Test: Placebo
- Cornea/Upper lid margin/Lower lid margin (Experimental): Subjects that are at least 18 years of age wearing their habitual lenses will be randomized into one of six unique sequences. For each region within a sequence, the two treatments will be randomly assigned to the left and right eye (anesthesia left eye/placebo right eye OR placebo left eye/anesthesia left eye).
  Interventions: Diagnostic Test: Local Anesthesia; Diagnostic Test: Placebo
- Cornea/Lower lid margin/Upper lid margin (Experimental): Subjects that are at least 18 years of age wearing their habitual lenses will be randomized into one of six unique sequences. For each region within a sequence, the two treatments will be randomly assigned to the left and right eye (anesthesia left eye/placebo right eye OR placebo left eye/anesthesia left eye).
  Interventions: Diagnostic Test: Local Anesthesia; Diagnostic Test: Placebo
- Upper lid margin/Cornea/Lower lid margin (Experimental): Subjects that are at least 18 years of age wearing their habitual lenses will be randomized into one of six unique sequences. For each region within a sequence, the two treatments will be randomly assigned to the left and right eye (anesthesia left eye/placebo right eye OR placebo left eye/anesthesia left eye).
  Interventions: Diagnostic Test: Local Anesthesia; Diagnostic Test: Placebo
- Lower lid margin/Upper lid margin/Cornea (Experimental): Subjects that are at least 18 years of age wearing their habitual lenses will be randomized into one of six unique sequences. For each region within a sequence, the two treatments will be randomly assigned to the left and right eye (anesthesia left eye/placebo right eye OR placebo left eye/anesthesia left eye).
  Interventions: Diagnostic Test: Local Anesthesia; Diagnostic Test: Placebo

INTERVENTIONS:
Diagnostic Test: Local Anesthesia — Minims Proxymetacaine hydrochloride Eye Drops
Diagnostic Test: Placebo — Sodium Chloride Solution

SUMMARY:
This is a controlled, randomized, subject-masked, 3x3 crossover, non-dispensing, contralateral study. Twenty subjects will be recruited based on their scores (with their habitual lenses) from the Contact Lens Dry Eye Questionnaire-8 and examined on four occasions.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. They are of legal age (18 years) and capacity of volunteer.
  2. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  3. They must appear able and willing to adhere to the instructions set forth in this clinical protocol.
  4. They have worn the same brand of soft spherical contact lenses for at least the previous three months, by self-report.
  5. They are defined as 'symptomatic' contact lens wearers (CLDEQ-8 score of 20-37) with their habitual contact lenses.
  6. They are willing to wear their lenses for approximately 14 hours on study days.
  7. They have a wearable pair of spectacles, if applicable.
  8. They agree not to participate in other clinical research for the duration of this study.
  9. They can attain high contrast logMAR visual acuity of 0.20 or better in their habitual contact lenses in each eye.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. They have an ocular disorder, which would normally contra-indicate contact lens wear.
  2. They have a systemic disorder, which would normally contra-indicate contact lens wear.
  3. They are using any topical medication such as eye drops or ointment.
  4. They have had cataract or corneal refractive surgery.
  5. They are pregnant or breast-feeding by self-report.
  6. They have any infectious disease (e.g. hepatitis) or any immunosuppressive disease (e.g. HIV), by self-report.
  7. They have any known hypersensitivity or allergic reaction to any of the known ingredients in the anesthetic.
  8. They have a history of severe allergic reaction or anaphylaxis.
  9. They have a history of cardiac disease or hyperthyroidism.
  10. They have taken part in any other contact lens or care solution clinical trial or research, within two weeks prior to starting this study.
  11. They are an employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  12. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
  13. They have grade 3 or greater of any of the following ocular surface signs which would contraindicate contact lens wear: corneal edema, corneal vascularisation, corneal staining, tarsal conjunctival changes or any other abnormality which would normally contraindicate contact lens wear.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 22 subjects were enrolled in this study. Of those enrolled, 20 were dispensed at least one study lens while 2 subjects failed to meet all eligibility criteria. Of those dispensed, 17 completed the study while 3 subjects were discontinued.
Groups:
- Lower Lid Margin/Upper Lid Margin/Cornea: Subjects assigned to recieved two treatmens contralaterally, in the lower lid margin during period 1, the upper lid margin during period 2 and the cornea at period 3.
- Lower Lid Margin/Cornea/Upper Lid Margin: Subjects assigned to recieved two treatmens contralaterally, in the lower lid margin during period 1, the cornea during period 2 and the upper lid margin during period 3.
- Upper Lid Margin/Lower Lid Margin/Cornea: Subjects assigned to recieved two treatmens contralaterally, in the upper lid margin during period 1, the lower lid margin during period 2 and the cornea during period 3.
- Upper Lid Margin/Cornea/Lower Lid Margin: Subjects assigned to recieved two treatmens contralaterally, in the upper lid margin during period 1, the cornea during period 2 and the lower lid margin during period 3.
- Cornea/Lower Lid Margin/Upper Lid Margin: Subjects assigned to recieved two treatmens contralaterally, in the Cornea during period 1, the lower lid margin during period 2 and the upper lid maring during period 3.
- Cornea/Upper Lid Margin/Lower Lid Margin: Subjects assigned to recieved two treatmens contralaterally, in the Cornea during period 1, the upper lid margin during period 2 and the lower lid maring during period 3.
Period: Period 1
Arm/Group | Lower Lid Margin/Upper Lid Margin/Cornea | Lower Lid Margin/Cornea/Upper Lid Margin | Upper Lid Margin/Lower Lid Margin/Cornea | Upper Lid Margin/Cornea/Lower Lid Margin | Cornea/Lower Lid Margin/Upper Lid Margin | Cornea/Upper Lid Margin/Lower Lid Margin
Started | 3 | 3 | 3 | 4 | 4 | 3
Completed | 3 | 3 | 3 | 4 | 4 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 2
Arm/Group | Lower Lid Margin/Upper Lid Margin/Cornea | Lower Lid Margin/Cornea/Upper Lid Margin | Upper Lid Margin/Lower Lid Margin/Cornea | Upper Lid Margin/Cornea/Lower Lid Margin | Cornea/Lower Lid Margin/Upper Lid Margin | Cornea/Upper Lid Margin/Lower Lid Margin
Started | 3 | 3 | 3 | 4 | 4 | 2
Completed | 3 | 2 | 3 | 4 | 4 | 2
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Unscuccessful Treatment | 0 | 1 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Lower Lid Margin/Upper Lid Margin/Cornea | Lower Lid Margin/Cornea/Upper Lid Margin | Upper Lid Margin/Lower Lid Margin/Cornea | Upper Lid Margin/Cornea/Lower Lid Margin | Cornea/Lower Lid Margin/Upper Lid Margin | Cornea/Upper Lid Margin/Lower Lid Margin
Started | 3 | 2 | 3 | 4 | 4 | 2
Completed | 2 | 2 | 3 | 4 | 4 | 2
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Dispensed Subjects: All subjects dispensed at least one study lens.
Arm/Group | All Dispensed Subjects
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.2 (70.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 3
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  Asian | 8
  Black or African Amercian | 2
  White | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 20

OUTCOME MEASURES:

1. Primary Outcome: Subjective Comfort Scores
Description: Subjects were asked to rate how comfortable each eye was overall using a visual analog scale of 0 to 100 where 0=worse comfort imaginable and 100=best comfort imaginable.
Time Frame: 5 and 10 Minutes post-treament
Population: All randomized subjects regardless of actual treatment and subsequent withdrawl from the study or deviation from protocol.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: eyes
Groups:
- Test (Anesthetic)- Cornea: Eyes that instilled the Test (Anesthetic) in either the right or left corneal ocular region.
- Placebo- Cornea: Eyes that instilled the Placebo in either the right or left corneal ocular region.
- Test (Anesthetic) - Upper Lid Margin: Eyes that instilled the Test in either the right or left upper lid margin.
- Placebo- Upper Lid Margin: Eyes that instilled the Placebo in either the right or left upper lid margin.
- Test (Anesthetic)- Lower Lid Margin: Eyes that instilled the Test in either the right or left lower lid margin.
- Placebo- Lower Lid Margin: Eyes that instilled the Placebo in either the right or left lower lid margin.
Arm/Group | Test (Anesthetic)- Cornea | Placebo- Cornea | Test (Anesthetic) - Upper Lid Margin | Placebo- Upper Lid Margin | Test (Anesthetic)- Lower Lid Margin | Placebo- Lower Lid Margin
Number analyzed (Participants) | 12 | 15 | 18 | 17 | 19 | 18
Number analyzed (eyes) | 12 | 15 | 18 | 17 | 19 | 18
Units on a Scale
  5- Mintues Post Treatment | 79.25 (8.925) | 70.93 (20.838) | 61.00 (20.807) | 61.94 (16.783) | 64.00 (20.915) | 61.06 (21.292)
  10- Mintues Post Treatment | 18.50 (10.265) | 72.33 (20.430) | 65.11 (21.766) | 64.00 (19.239) | 70.79 (16.511) | 63.17 (20.667)
Statistical Analysis 1: Comparison: Test (Anesthetic)- Cornea vs Placebo- Cornea; 5-Mintues Post Treatment; Test type: Superiority — Subjective comfort was analyzed using linear mixed model. Statistical inference was made based on the 95% confidence interval constructed for the least square mean difference; Linear Mixed Model; Least-Square Mean Difference = 2.6, 95% CI 2-sided [-7.3 to 12.4], Standard Error of Mean 4.96 — Difference was calculated as Test - Placebo
Statistical Analysis 2: Comparison: Test (Anesthetic)- Cornea vs Placebo- Cornea; 10-Minutes Post Treatment; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Least-square Mean Difference = 0.9, 95% CI 2-sided [-9.6 to 11.5], Standard Error of Mean 5.30 — Difference was calculated as Test - Placebo
Statistical Analysis 3: Comparison: Test (Anesthetic) - Upper Lid Margin vs Placebo- Upper Lid Margin; 5-Minutes Post Treatment; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Least-Square Mean Difference = 0.8, 95% CI 2-sided [-8.2 to 9.8], Standard Error of Mean 4.67 — difference was calculated as Test - Placebo
Statistical Analysis 4: Comparison: Test (Anesthetic) - Upper Lid Margin vs Placebo- Upper Lid Margin; 10-Mintues Post Treatment; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Least-square Mean Difference = 2.9, 95% CI 2-sided [-6.5 to 12.2], Standard Error of Mean 4.67 — Difference was calculated as Test - Placebo
Statistical Analysis 5: Comparison: Test (Anesthetic)- Lower Lid Margin vs Placebo- Lower Lid Margin; 5-Mintues Post Treatment; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Least-square Mean Difference = 3.0, 95% CI 2-sided [-5.7 to 11.7], Standard Error of Mean 4.37 — Difference was calculated as Test - Placebo
Statistical Analysis 6: Comparison: Test (Anesthetic)- Lower Lid Margin vs Placebo- Lower Lid Margin; 10-Mintues Post Treatment; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Least-sqaure Mean Difference = 7.7, 95% CI 2-sided [-1.4 to 16.8], Standard Error of Mean 4.54 — difference was calculated as Test - Placebo

2. Primary Outcome: Change in Subjective Comfort Scores From Pre-treatment to Post-treatment
Description: Subjects were asked to rate how comfortable each eye was overall using a visual analog scale of 0 to 100 where 0=worse comfort imaginable and 100=best comfort imaginable. Subjects wore their habitual contacts during the pre-treatment assessment.
Time Frame: 14-Hours upon Lens-Insertion (pre-treatment), and 10 Minutes post-treament
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: eyes
Arm/Group | Test (Anesthetic)- Cornea | Placebo- Cornea | Test (Anesthetic) - Upper Lid Margin | Placebo- Upper Lid Margin | Test (Anesthetic)- Lower Lid Margin | Placebo- Lower Lid Margin
Number analyzed (Participants) | 12 | 15 | 18 | 17 | 19 | 18
Number analyzed (eyes) | 12 | 15 | 18 | 17 | 19 | 18
Units on a Scale
  5- Mintues Post Treatment | 79.25 (8.925) | 70.93 (20.838) | 61.00 (20.807) | 61.94 (16.783) | 64.00 (20.915) | 61.06 (21.292)
  10- Mintues Post Treatment | 18.50 (10.265) | 72.33 (20.430) | 65.11 (21.766) | 64.00 (19.239) | 70.79 (16.511) | 63.17 (20.667)
  Pre-treatment | 62.35 (23.238) | 60.16 (24.862) | 56.67 (24.867) | 58.35 (24.746) | 60.11 (24.669) | 57.94 (21.939)
Statistical Analysis 1: Comparison: Test (Anesthetic)- Cornea vs Placebo- Cornea; 5-Mintues Post Treatment; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Least-Square Mean Difference = 2.1, 95% CI 2-sided [-10.3 to 14.4], Standard Error of Mean 6.22 — Difference was calculated as Test - Placebo
Statistical Analysis 2: Comparison: Test (Anesthetic)- Cornea vs Placebo- Cornea; 10-Minutes Post Treatment; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Least-square Mean Difference = 0.4, 95% CI 2-sided [-12.1 to 12.9], Standard Error of Mean 6.30 — Difference was calculated as Test - Placebo
Statistical Analysis 3: Comparison: Test (Anesthetic) - Upper Lid Margin vs Placebo- Upper Lid Margin; 5-Minutes Post Treatment; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Least-Square Mean Difference = 0.3, 95% CI 2-sided [-11.4 to 12.1], Standard Error of Mean 5.92 — difference was calculated as Test - Placebo
Statistical Analysis 4: Comparison: Test (Anesthetic) - Upper Lid Margin vs Placebo- Upper Lid Margin; 10-Mintues Post Treatment; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Least-square Mean Difference = 2.4, 95% CI 2-sided [-9.2 to 14.0], Standard Error of Mean 5.83 — Difference was calculated as Test - Placebo
Statistical Analysis 5: Comparison: Test (Anesthetic)- Lower Lid Margin vs Placebo- Lower Lid Margin; 5-Mintues Post Treatment; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Least-square Mean Difference = 2.9, 95% CI 2-sided [-8.5 to 14.3], Standard Error of Mean 5.76 — Difference was calculated as Test - Placebo
Statistical Analysis 6: Comparison: Test (Anesthetic)- Lower Lid Margin vs Placebo- Lower Lid Margin; 10-Mintues Post Treatment; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Least-sqaure Mean Difference = 7.6, 95% CI 2-sided [-3.7 to 18.8], Standard Error of Mean 5.67 — difference was calculated as Test - Placebo

3. Primary Outcome: Subjective Comfort Score Difference Between Post-treatment and Post-insertion Within Anesthetic
Description: Subjects were asked to rate how comfortable each eye was overall on the scale of 0 to 100 where 0=worse comfort imaginable and 100=best comfort imaginable.
Time Frame: Immediately after lens-insertion, 5 and 10 minutes post-treatment
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: eyes
Groups:
- Test (Anesthetic)- Corneal: Eyes that instilled the Test (Anesthetic) in either the right or left corneal ocular region.
Arm/Group | Test (Anesthetic)- Corneal | Test (Anesthetic) - Upper Lid Margin | Test (Anesthetic)- Lower Lid Margin
Number analyzed (Participants) | 12 | 18 | 19
Number analyzed (eyes) | 12 | 18 | 19
Units on a Scale
  Immediate Post Lens Insertion | 78.06 (17.243) | 73.33 (22.646) | 80.37 (14.064)
  5-Minutes Post Treatment | 79.25 (8.925) | 61.00 (20.807) | 64.00 (20.915)
  10 Minutes Post Treatment | 78.50 (10.265) | 65.11 (21.766) | 70.79 (16.511)
Statistical Analysis 1: Comparison: Test (Anesthetic)- Corneal; 5-Minutes Post Treatment; Test type: Superiority — Superiority was concluded if the lower limit of 95% confidence interval was greater than 0 for at least one of the three ocular regions (upper lid margin, lower lid margin, or cornea); Mixed Models Analysis; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-13.2 to 5.1], Standard Error of Mean 4.61; Mean difference was calculated as (5-min Post-Treatment MINUS Immediate Post-insertion)
Statistical Analysis 2: Comparison: Test (Anesthetic)- Corneal; 10-Minutes Post Treatment; Test type: Superiority — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-13.9 to 5.3], Standard Error of Mean 4.85; Mean difference was calculated as (10-min Post-Treatment MINUS Immediate Post-insertion)
Statistical Analysis 3: Comparison: Test (Anesthetic)- Lower Lid Margin; 5-Minutes Post Treatment; Test type: Superiority — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = -16.4, 95% CI 2-sided [-24.4 to -8.3], Standard Error of Mean 4.04; Mean difference was calculated as (5-min Post-Treatment MINUS Immediate Post-insertion)
Statistical Analysis 4: Comparison: Test (Anesthetic)- Lower Lid Margin; 10-Minutes Post Treatment; Test type: Superiority — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = -9.6, 95% CI 2-sided [-17.8 to -1.4], Standard Error of Mean 4.14; Mean difference was calculated as (10-min Post-Treatment MINUS Immediate Post-insertion)
Statistical Analysis 5: Comparison: Test (Anesthetic) - Upper Lid Margin; 5-Minutes Post Treatment; Test type: Superiority — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = -12.3, 95% CI 2-sided [-20.6 to -4.1], Standard Error of Mean 4.15; Mean difference was calculated as (5-min Post-Treatment MINUS Immediate Post-insertion)
Statistical Analysis 6: Comparison: Test (Anesthetic) - Upper Lid Margin; 10-Minutes Post Treatment; Test type: Superiority — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = -8.2, 95% CI 2-sided [-16.7 to 0.2], Standard Error of Mean 4.25; Mean difference was calculated as (10-min Post-Treatment MINUS Immediate Post-insertion)

4. Secondary Outcome: Change in Subjective Comfort Between Ocular Regions at Posttreatment Within Anesthetic
Description: as for outcome 3
Time Frame: 5 and 10 minutes post treatment
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: eyes
Arm/Group | Test (Anesthetic)- Corneal | Test (Anesthetic) - Upper Lid Margin | Test (Anesthetic)- Lower Lid Margin
Number analyzed (Participants) | 12 | 18 | 19
Number analyzed (eyes) | 12 | 18 | 19
Units on a Scale
  5-Minutes Post Treatment | 79.25 (8.925) | 61.00 (20.807) | 64.00 (20.915)
  10 Minutes Post Treatment | 78.50 (10.265) | 65.11 (21.766) | 70.79 (16.511)
Statistical Analysis 1: Comparison: Test (Anesthetic)- Corneal vs Test (Anesthetic)- Lower Lid Margin; 10-Minutes Post Treatment; Test type: Superiority — Superiority was concluded if the lower limit of 95% confidence interval was greater than 0; Mixed Models Analysis; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-8.7 to 11.6], Standard Error of Mean 5.07; Mean Difference was cacluated as Corneal - Lower Lid Margin
Statistical Analysis 2: Comparison: Test (Anesthetic)- Corneal vs Test (Anesthetic)- Lower Lid Margin; 5-Minutes Post Treatment; Test type: Superiority — Superiority was concluded if the lower limit of 95% confidence interval was greater than 0; Mixed Models Analysis; Mean Difference (Final Values) = 8.5, 95% CI 2-sided [-1.0 to 18.0], Standard Error of Mean 4.77; Mean Difference was cacluated as Corneal - Lower Lid Margin
Statistical Analysis 3: Comparison: Test (Anesthetic)- Corneal vs Test (Anesthetic) - Upper Lid Margin; 10-Minutes Post Treatment; Test type: Superiority — Superiority was concluded if the lower limit of 95% confidence interval was greater than 0; Mixed Models Analysis; Mean Difference (Final Values) = 6.8, 95% CI 2-sided [-3.5 to 17.0], Standard Error of Mean 5.12; Mean Difference was cacluated as Corneal - Upper Lid Margin
Statistical Analysis 4: Comparison: Test (Anesthetic)- Corneal vs Test (Anesthetic) - Upper Lid Margin; 5-Minutes Post Treatment; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = 11.2, 95% CI 2-sided [1.6 to 20.8], Standard Error of Mean 4.82; Mean Difference was cacluated as Corneal - Upper Lid Margin

5. Secondary Outcome: Change in Subjective Comfort From Pre-treatment to Post-Treatment Between Ocular Regions
Description: as for outcome 3
Time Frame: 14 hours upon lens-insertion (pre-treatment), 5- and 10- minutes post-treatment
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: eyes
Arm/Group | Test (Anesthetic)- Corneal | Test (Anesthetic) - Upper Lid Margin | Test (Anesthetic)- Lower Lid Margin
Number analyzed (Participants) | 12 | 18 | 19
Number analyzed (eyes) | 12 | 18 | 19
Units on a Scale
  Pre-Treatment | 62.35 (23.238) | 56.67 (24.867) | 60.16 (24.862)
  5-Minutes Post Treatment | 79.25 (8.925) | 61.00 (20.807) | 64.00 (20.915)
  10-Minutes Post Treatment | 78.50 (10.265) | 65.11 (21.766) | 70.79 (16.511)
Statistical Analysis 1: Comparison: Test (Anesthetic)- Corneal vs Test (Anesthetic)- Lower Lid Margin; 10-Minutes Post Treatment; Test type: Superiority — Superiority was concluded if the lower limit of 95% confidence interval was greater than 0; Mixed Models Analysis; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-11.4 to 12.9], Standard Error of Mean 6.12; Mean Difference was cacluated as Corneal - Lower Lid Margin: 10-mintues post treatment - Pre Treatment
Statistical Analysis 2: Comparison: Test (Anesthetic)- Corneal vs Test (Anesthetic)- Lower Lid Margin; 5-Minutes Post Treatment; Test type: Superiority — Superiority was concluded if the lower limit of 95% confidence interval was greater than 0; Mixed Models Analysis; Mean Difference (Final Values) = 7.8, 95% CI 2-sided [-4.9 to 19.9], Standard Error of Mean 6.10; Mean Difference was cacluated as Corneal - Lower Lid Margin: 5-mintues post treatment - Pre Treatment
Statistical Analysis 3: Comparison: Test (Anesthetic)- Corneal vs Test (Anesthetic) - Upper Lid Margin; 10-Minutes Post Treatment; Test type: Superiority — Superiority was concluded if the lower limit of 95% confidence interval was greater than 0; Mixed Models Analysis; Mean Difference (Final Values) = 2.9, 95% CI 2-sided [-9.3 to 15.2], Standard Error of Mean 6.19; Mean Difference was cacluated as Corneal - Upper Lid Margin: 10-mintues post treatment - Pre Treatment
Statistical Analysis 4: Comparison: Test (Anesthetic)- Corneal vs Test (Anesthetic) - Upper Lid Margin; 5-Minutes Post Treatment; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Final Values) = 7.4, 95% CI 2-sided [-4.9 to 19.6], Standard Error of Mean 6.17; Mean Difference was cacluated as Corneal - Upper Lid Margin: 5-mintues post treatment - Pre Treatment

6. Secondary Outcome: Subjective Comfort Difference Between Post-removal and Preinsertion Within Anesthetic and Cornea
Description: as for outcome 3
Time Frame: Immediately before lens-insertion (pre-insertion), 30 seconds after lens removal
Population: All randomized subjects regardless of actual treatment and subsequent withdrawl from study or deviation from protocol.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Eyes
Arm/Group | Test (Anesthetic)- Cornea
Number analyzed (Participants) | 12
Number analyzed (Eyes) | 12
Units on a Scale
  Pre-Insertion | 81.53 (17.784)
  Post-Removal | 69.12 (21.508)
Statistical Analysis 1: Comparison: Test (Anesthetic)- Cornea; Test type: Superiority — Superiority was concluded if the lower limit of 95% confidence interval was greater than 0; Mixed Models Analysis; Mean Difference (Final Values) = -12.4, 95% CI 2-sided [-20.9 to -3.9], Standard Error of Mean 4.22; mean difference was calculated as postremoval minus pre-insertion with Test and corneal region

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Up to 6-weeks per subject.
Groups:
- Placebo: subjects that were exposed to the placebo during any point in the study.
- Test (Anesthetic): Subjects that were exposed to the Anesthetic during any point in the study.
Arm/Group | Placebo | Test (Anesthetic)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT03733899/Prot_SAP_000.pdf